CLINICAL TRIAL: NCT03228316
Title: Superior Hypogastric Plexus Block and Pulsed Radiofrequency on Dorsal Root Ganglia of Sacral Nerves for Chronic Pelvic Cancer Pain
Brief Title: Superior Hypogastric Plexus Block Versus Pulsed Radiofrequency for Chronic Pelvic Cancer Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, marina emeel helal, principle invistigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MEHG
Record Dates: First submitted 2017-06-15; First posted 2017-07-24 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-07

CONDITIONS: Chronic Pelvic Cancer Pain
MeSH Terms: interventions — Pulsed Radiofrequency Treatment

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: prospective interventional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the study group one (Experimental): 20 patients with superior hypogastric plexus block
  Interventions: Procedure: superior hypogastric plexus block
- the study group two (Experimental): 20 patients with superior hypogastric plexus block combined to pulsed radiofrequency on sacral nerve roots 2,3 and 4
  Interventions: Procedure: superior hypogastric plexus block; Radiation: pulsed radiofrequency

INTERVENTIONS:
Procedure: superior hypogastric plexus block — nerve plexus block
Radiation: pulsed radiofrequency — pulsed radiofrequency on sacral nerve roots 2,3 and 4
  Arms: the study group two

SUMMARY:
Cancer-related pain represents a major challenge for both clinicians and patients. This pain can be associated directly with the cancer or with certain treatments administered to the patient. 52.1% of cancer patients suffer from pain and that 62.6% are not satisfied with the current pain treatment. Pain prevalence is high in developing countries due to late diagnosis and major impediments to opioid access

DETAILED DESCRIPTION:
pelvic cancer is a broad term encompassing malignant tumors of the bladder, prostate, cervix, endometrium, ovaries, and uterus, among others. Pain associated with pelvic cancer is one of the most debilitating symptoms experienced by affected patients. Multiple studies demonstrate that the prevalence of pain in patients with pelvic cancer is >50%, and can be upwards of 60% to 70% in patients with advanced or metastatic disease . Cancer patients with extension of tumor into the pelvis may experience severe pain. Oral or parenteral opioids may not only fail to provide relief, but may cause excessive sedation and other side effects. More invasive approaches may thus be needed to control pain and improve the quality of life. Since pelvic cancer pain is visceral in most cases, this could be achieved with percutaneous chemical neurolytic block of the superior hypogastric plexus . The superior hypogastric plexus is located at the anterior aspect of the L5 and S1 vertebrae, and traverses the disk between these levels. It is an extension of the aortic plexus below the aortic bifurcation, and contains almost exclusively sympathetic ﬁbers and visceral afferents . Afferent pain ﬁbers innervating pelvic organs travel with sympathetic nerves, trunks, ganglia, and rami; thus, interrupting the sympathetic chain at this level can be used to treat pelvic cancer pain. Several studies examined the use of superior hypogastric plexus block in the treatment of pelvic cancer pain. Although the authors reported a mean reduction in pain of 70%, neither the follow-up period nor the proportion with a successful prognostic block were noted. Radiofrequency utilizes a high-frequency alternating current that is passed from the needle electrode into the surrounding tissue, resulting in frictional heating and necrosis. Due to the accuracy of lesions produced by radiofrequency ablation, there has been growing interest in the use of this technique for neurolysis of nerves as it offers the potential of accurate nerve destruction ablation, with a predictable and controlled ablative lesion. Another advantage of radiofrequency ablation is that it has an immediate effect unlike alcohol and phenol, which may take up to 1 week or 10 days to achieve neurolysis .

ELIGIBILITY:
Inclusion Criteria:

* sympathetically maintained pelvic, perineal pain
* pain is no longer controlled with oral morphine sustained release tablets 30 mg
* excessive sedation or other side effects from oral morphine sustained release tablets 30 mg or amitryptyline tablets 25 mg
* age between 18-70 years

Exclusion Criteria:

* patient refusal
* patients with coagulopathies
* allergy to constant dyes or phenol
* patients receiving radiation or chemotherapy within 4 weeks of neurolytic block
* patients with major or moderate cardiac/respiratory incapacitating diseases
* liver and renal failure
* patients younger than 18 years and older than 70 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-10-20 (Estimated); Primary Completion 2020-06-20 (Estimated); Study Completion 2020-12-20 (Estimated)

PRIMARY OUTCOMES:
Visual analogue score for pain | 2 months
  Points on a scale

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sindt JE, Brogan SE. Interventional Treatments of Cancer Pain. Anesthesiol Clin. 2016 Jun;34(2):317-39. doi: 10.1016/j.anclin.2016.01.004. PMID 27208713
- [Derived] Hetta DF, Mohamed AA, Abdel Eman RM, Abd El Aal FA, Helal ME. Pulsed Radiofrequency of the Sacral Roots Improves the Success Rate of Superior Hypogastric Plexus Neurolysis in Controlling Pelvic and Perineal Cancer Pain. Pain Physician. 2020 Mar;23(2):149-157. PMID 32214294
- Available data/document: Clinical Study Report — http://www.ncbi.nlm.nih.gov/pubmed/27208713